CLINICAL TRIAL: NCT00299728
Title: A Phase I Study Using Vaccination With NY-ESO-1 Recombinant Protein Mixed With CpG 7909 and Montanide ISA-51 VG in Patients With Cancers That Often Express NY-ESO-1.
Brief Title: NY-ESO-1 Protein With Montanide and CpG 7909 as Cancer Vaccine in Several Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2003-022;NYU05-120;CUMC9147
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Tumors
Keywords: NY-ESO-1; Vaccine; Adjuvant or metastatic setting; Several tumor types eligible
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A; 100 μg NY-ESO-1 protein co-mixed with CpG 7909 and Montanide ISA-51 VG (Experimental): 100 μg NY-ESO-1 protein co-mixed with 2.5 mg CpG 7909 and 1.25 mL Montanide ISA-51 VG. The vaccine was administered subcutaneously every 3 weeks for a total of 4 doses (study weeks 1, 4, 7 and 10).
  Interventions: Biological: NY-ESO-1 Protein Vaccine
- Arm B; 400 μg NY-ESO-1 protein co-mixed with CpG 7909 and Montanide ISA-51 VG (Experimental): 400 μg NY-ESO-1 protein co-mixed with 2.5 mg CpG 7909 and 1.25 mL Montanide ISA-51 VG. The vaccine was administered subcutaneously every 3 weeks for a total of 4 doses (study weeks 1, 4, 7 and 10).
  Interventions: Biological: NY-ESO-1 Protein Vaccine

INTERVENTIONS:
Biological: NY-ESO-1 Protein Vaccine — NY-ESO-1 recombinant protein mixed with CpG 7909 and Montanide ISA-51 VG

SUMMARY:
This is a Phase I, open-label, randomized study of NY-ESO-l protein with immune adjuvants CpG 7909 and Montanide ISA-51 VG in patients with tumors that often express NY-ESO-1.

The vaccinations was to be administered subcutaneously every 3 weeks for 4 doses.

Patients with any malignancy that is known to frequently express NY-ESO-1 were eligible, regardless of whether antigen expression in the autologous tumor could be demonstrated or not by either PCR or immunohistochemistry.

The primary objective of the study was to define safety.

Secondarily, the study was to evaluate whether patients developed a specific immunologic response to the NY-ESO-1 protein. Blood samples were to be obtained at baseline, prior to each vaccination, one week after each vaccination, and at the last study visit for the assessment of NY-ESO-1-specific CD4+ and CD8+ T cells. Cytokine secretion by NY-ESO-1-specific CD8+ and CD4+ T cells, as a measure of T cell activation, was to be determined by FACS analysis. In addition, humoral immunity was to be determined by the presence of NY-ESO-1-specific antibodies which were to be assessed in all patients by ELISA.

Disease status was to be assessed at baseline and 2-4 weeks after the fourth vaccination in patients with evaluable (measurable and non-measurable) disease.

DETAILED DESCRIPTION:
Subjects were to receive an investigational (research) cancer vaccine every 3 weeks for a total of 4 treatments. It was given by injection underneath the skin in an extremity (leg or arm). A vaccine is a compound designed to strengthen the immune system (the cells and substances that protect the body from infection and foreign matter) to fight an illness such as infections or cancer. This vaccine is called NY-ESO-1 protein. NY-ESO-1 protein (an antigen, which is a compound that is recognized by the immune system) is found in many cancers. Proteins such as NY-ESO-1 and their fragments are the targets the immune system needs to recognize cancer cells. If the immune system can recognize these antigens (foreign substances) it may be able to kill the cells that carry them. NY-ESO-1 can be found at different stages of cancers, and is likely to be expressed (shown) at some point in the lifecycle of these types of cancer (that are eligible for this study). Therefore this study tries to boost (strengthen) the immune system toward NY-ESO-1 protein regardless of whether it is found in your tumor or not.

Since we do not know whether different doses of the NY-ESO-1 protein may result in varying degrees of immune stimulation, we will be randomizing (that is, at the flip of a coin or, in other words, by chance). You may receive either the lower dose of NY-ESO-1 protein (100 µg) or the higher dose (400 µg).

The NY-ESO-1 protein vaccine was to be mixed with 2 substances, called adjuvants (the full names are: CPG 7909 and Montanide ISA-51 VG). Adjuvants are substances to increase the vaccine's ability to stimulate the immune system. By adding two adjuvants to the vaccine, it is hoped that the boosting of the immune system will be especially effective.

It is important to understand, that vaccines are only experimental (investigational, research) for the treatment of cancer. They are not approved by the Food and Drug Administration (FDA) as treatment. Therefore they are only offered in clinical trials.

All tests and treatments were performed as an outpatient.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of hepatocellular carcinoma, bladder cancer, breast cancer, non-small lung cancer (NSCLC), melanoma, sarcoma, prostate cancer, esophageal cancer, or ovarian cancer, independent of NY-ESO-1 expression in a tumor biopsy.

   or

   Histological diagnosis of other types of cancers, provided NY-ESO-1 or LAGE-1 expression can be shown in a tumor biopsy.
2. At least 4 weeks since surgery prior to first dosing of study agent.
3. Laboratory values within the following limits:

   * Hemoglobin ≥ 11.0 g/dL
   * Neutrophil count ≥ 1.5 x l0^9/L
   * Lymphocyte count ≥ lower limit of institutional normal
   * Platelet count ≥ 80 x l0^9/L
   * Serum creatinine ≤ 2.0 mg/dL
   * Serum bilirubin ≤ 2 x upper limit of institutional normal
   * AST/ALT ≤ 2 x upper limit of institutional normal
4. Patients must have a Karnofsky performance status of ≥70%.
5. Life expectancy ≥ 6 months.
6. Age ≥ 18 years.
7. Able and willing to give witnessed, written informed consent for participation in the trial.

Exclusion Criteria:

1. Clinically significant heart disease (i.e. NYHA class 3 congestive heart failure; myocardial infarction within the past six months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
2. Other serious illnesses, eg, serious infections requiring antibiotics, bleeding disorders.
3. Previous bone marrow or stem cell transplant.
4. History of immunodeficiency disease or autoimmune disease except vitiligo.
5. Metastatic disease to the central nervous system, unless treated and stable.
6. Other malignancy within 3 years prior to entry into the study, except for treated early-stage melanoma or non-melanoma skin cancer, or cervical carcinoma in situ.
7. Known HIV, Hepatitis B or Hepatitis C positivity.
8. Chemotherapy, radiation therapy or immunotherapy within 4 weeks prior to first dose of study agent (6 weeks for nitrosoureas).
9. Concomitant treatment with steroids. Topical or inhalational steroids are permitted.
10. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dose of study agent.
11. Pregnancy or lactation.
12. Women of childbearing potential not using a medically acceptable means of contraception.
13. Psychiatric or addictive disorders that may compromise the ability to give informed consent.
14. Lack of availability of the patient for immunological and clinical follow-up assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-03-21 (Actual); Primary Completion 2006-10-10 (Actual); Study Completion 2014-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — NYU Langone Health; Sylvia Adams, MD, Study Director — NYU Langone Health; Gregory Mears, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - NYU Clinical Cancer Center, New York, New York
  - NY Presbyterian- Columbia, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Valmori D, Souleimanian NE, Tosello V, Bhardwaj N, Adams S, O'Neill D, Pavlick A, Escalon JB, Cruz CM, Angiulli A, Angiulli F, Mears G, Vogel SM, Pan L, Jungbluth AA, Hoffmann EW, Venhaus R, Ritter G, Old LJ, Ayyoub M. Vaccination with NY-ESO-1 protein and CpG in Montanide induces integrated antibody/Th1 responses and CD8 T cells through cross-priming. Proc Natl Acad Sci U S A. 2007 May 22;104(21):8947-52. doi: 10.1073/pnas.0703395104. Epub 2007 May 15. PMID 17517626

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A; 100 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG | Arm B; 400 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG
Started | 11 | 11
Completed | 11 | 8
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Progressive disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who entered the study and received the NY-ESO-1 protein vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A; 100 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG | Arm B; 400 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (15.5) | 56 (12.7) | 54.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Adverse Events (AEs) and Dose-limiting Toxicities (DLTs)
Description: All AEs occurring during the study were documented in the source records and on the respective AE case report form (CRF) pages, regardless of the assumption of a causal relationship. All events that occurred after the first administration of study drug were to be documented. The severity of an AE was assessed according to the NCI CTCAE scale (Version 3.0).
  DLT was defined as ≥ Grade 3 hematological and non-hematological toxicities or ≥ Grade 2 allergic reaction for generalized urticaria that was definitely, probably, or possibly related to the administration of the NY-ESO-1 protein vaccine.
Time Frame: up to 14 weeks
Population: All subjects who entered the study and received the NY-ESO-1 protein vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A; 100 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG | Arm B; 400 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG
Number analyzed (Participants) | 11 | 11
Participants
  Number of subjects reporting AEs | 11 | 11
  Number of subjects with DLTs | 0 | 0

2. Primary Outcome: Number of Subjects With NY-ESO-1-Specific Humoral Immunity as Determined by an Increase in Antibody Titer From Baseline.
Description: Blood samples were taken at baseline and in weeks 2, 4, 5, 7, 8, 10, 11, and 12-14 for the assessment of NY-ESO-1-specific antibodies by an enzyme-linked immunosorbent assay (ELISA). Sera were assessed over a range of dilutions from 1/100 to 1/100,000. Titers were calculated as the serum dilution giving 50% of maximal optical density obtained by using a standard positive serum. Positive results were reciprocal serum titers greater than 100.
Time Frame: Up to 14 weeks
Population: All subjects who entered the study and received the NY-ESO-1 protein vaccine and had antibody titers measured both pre-and post-treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A; 100 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG | Arm B; 400 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG
Number analyzed (Participants) | 11 | 7
Participants
  Number of subjects with positive antibody titers at baseline and after treatment | 1 | 0
  Number of subjects with negative titers at baseline and positive titers following treatment | 10 | 7

3. Secondary Outcome: Number of Subjects With Tumor Responses as Measured by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Computed tomography (CT) or magnetic resonance imaging (MRI) scans were performed at screening and weeks 12-14 and 16-18, and tumor response was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) according to Therasse P et al. 2000.
  Per RECIST, target lesions were categorized as follows: complete response (CR): disappearance of all target lesions; partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria; no evidence of disease (NED): no evidence of disease at baseline and post-baseline assessments.
Time Frame: up to 18 weeks
Population: All subjects who entered the study and received the NY-ESO-1 protein vaccine and had at least one post-treatment tumor assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A; 100 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG | Arm B; 400 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG
Number analyzed (Participants) | 11 | 10
Participants
  CR | 0 | 0
  PR | 0 | 0
  SD | 2 | 0
  PD | 0 | 2
  NED | 9 | 8

4. Secondary Outcome: Number of Subjects With NY-ESO-1 Specific Cellular Immunity as Measured by an Increase in NY-ESO-1-Specific CD4+ T Cells After in Vitro Stimulation
Description: Blood samples were taken at baseline and in weeks 2, 4, 5, 7, 8, 10, 11, 12-14, 16-18, 20-22, 24-26, and 28-32. Subjects were consented separately for blood draws after week 14. The induction of specific T cells was assessed after in vitro stimulation of pre- and post-treatment samples with a pool of overlapping peptides spanning the protein sequence, followed by quantification of specific IFN-γ-producing cells by intracellular staining. The response was considered significant if the frequency of T cells detected in at least one post-treatment sample exceeded by 3-fold that found in the baseline sample.
Time Frame: up to 32 weeks
Population: All subjects who entered the study, received the NY-ESO-1 protein vaccine and had pre- and post-treatment samples analyzed for NY-ESO-1 Specific CD4+ T cells.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A; 100 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG | Arm B; 400 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG
Number analyzed (Participants) | 11 | 7
Participants
  Number of subjects with an increase of NY-ESO-1 Specific CD4+ T cells after treatment | 10 | 7
  Number of subjects without an increase of NY-ESO-1 Specific CD4+ T cells after treatment | 1 | 0

5. Secondary Outcome: Number of Subjects With NY-ESO-1-Specific Cellular Immunity as Measured by an Increase in NY-ESO--Specific CD8+ T Cells After in Vitro Stimulation
Description: as for outcome 4
Time Frame: up to 32 weeks
Population: All subjects who entered the study, received the NY-ESO-1 protein vaccine and had pre- and post-treatment samples analyzed for NY-ESO-1-Specific CD8+ T cells.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A; 100 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG | Arm B; 400 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG
Number analyzed (Participants) | 11 | 7
Participants
  Number of subjects with an increase of NY-ESO-1-Specific CD8+ T cells after treatment | 5 | 4
  Number of subjects without an increase of NY-ESO-1-Specific CD8+ T cells after treatment | 6 | 3

ADVERSE EVENTS:
Time Frame: up to 14 weeks
Description: All AEs occurring during the study were documented in the source records and on the respective AE case report form (CRF) pages, regardless of the assumption of a causal relationship. All events that occurred after the first administration of study drug up to the end of week 14 were to be documented. The severity of an AE was assessed according to the NCI CTCAE scale (Version 3.0).
Arm/Group | Arm A; 100 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG | Arm B; 400 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 11/11 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A; 100 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG (N=11) | Arm B; 400 μg NY-ESO-1 Protein Co-mixed With CpG 7909 and Montanide ISA-51 VG (N=11)
Injection site induration (General disorders) | 11 | 9
Injection site erythema (General disorders) | 8 | 8
Injection site discomfort (General disorders) | 7 | 6
Injection site pain (General disorders) | 5 | 8
Fatigue (General disorders) | 6 | 6
Injection site nodule (General disorders) | 6 | 5
Injection site pruritus (General disorders) | 3 | 3
Injection site reaction (General disorders) | 3 | 2
Pyrexia (General disorders) | 7 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Headache (Nervous system disorders) | 6 | 2
Edema peripheral (General disorders) | 2 | 2
Body temperature increased (Investigations) | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Induration (General disorders) | 1 | 1
Injection site haematoma (General disorders) | 2 | 0
Injection site swelling (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Injection site discoloration (General disorders) | 0 | 1
Injection site injury (General disorders) | 0 | 1
Injection site rash (General disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Migrane (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No